CLINICAL TRIAL: NCT07279259
Title: Thrombolysis in Early Acute Ischemic Stroke Trial-Blood Pressure Management, EAST-BP
Brief Title: Thrombolysis in Early Acute Ischemic Stroke Trial-Blood Pressure Management
Acronym: EAST-BP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai 7th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAST-BP
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Acute Ischemic Stroke; Thrombolysis
Keywords: acute ischemic stroke; blood pressure; thrombolysis
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: central randomization with stratification
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor is independent of the treatment team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual BP management group (Other)
  Interventions: Procedure: Usual BP management group
- Adjusted BP management group (Experimental)
  Interventions: Procedure: Adjusted BP management group

INTERVENTIONS:
Procedure: Adjusted BP management group — For patients intended to receive intravenous thrombolysis, when the blood pressure ranges from 180/100 mmHg to 200/110 mmHg, simultaneous initiation of both intravenous thrombolysis and antihypertensive treatment can be considered. If the blood pressure exceeds 200/110 mmHg, antihypertensive treatment should be initiated first. Intravenous thrombolysis can be commenced after the blood pressure is reduced to below 200/110 mmHg. Before thrombolysis and within 24 hours after the initiation of intravenous thrombolysis, efforts should be made to control the extent of blood pressure reduction. When the blood pressure drops below 180/100 mmHg, antihypertensive treatment should be terminated. Twenty-four hours later, the routine blood pressure management protocol should be reinstated.
  Arms: Adjusted BP management group
Procedure: Usual BP management group — To receive blood pressure management according to standard local guidelines. In China, for patients scheduled for intravenous thrombolysis who present with elevated blood pressure, it is advised to maintain blood pressure below 180/100 mmHg for 24 hours, after which standard guideline-based blood pressure management should be resumed.
  Arms: Usual BP management group

SUMMARY:
This study is a Phase II, exploratory, prospective, multicenter, open-label, randomized controlled clinical trial with blinded endpoint assessment setting on the safety of an adjusted versus a conventional blood pressure management strategy during intravenous thrombolysis in AIS patients, with a key focus on the incidence of symptomatic intracranial hemorrhage (sICH).

DETAILED DESCRIPTION:
This study is a Phase II, exploratory, prospective, multicenter, open-label, randomized controlled clinical trial with blinded endpoint assessment. EAST-BP aims to investigate the safety of an adjusted versus a conventional blood pressure management strategy during intravenous thrombolysis in AIS patients, according to an ordinal analysis of Proportion of symptomatic intracranial hemorrhage within 24 hours after thrombolysis, proportion of severe or life-threatening major hemorrhage, DNT time for intravenous thrombolysis patients, proportion of independent functional prognosis at 90 days (90-day mRS 0-2), sequential analysis of improved 90-day mRS score for patients, proportion of death at 90 days, and neurological function status at 7 days or at discharge (if hospital stay is less than 7 days) .

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years (inclusive);
2. Patients with acute ischemic stroke;
3. Planned to receive intravenous thrombolysis within 4.5 hours of onset;
4. Elevated blood pressure: Before receiving intravenous thrombolysis treatment, blood pressure is elevated: systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg (defined as two consecutive measurements within 2 minutes);
5. Informed consent signed (or signed by a proxy).

Exclusion Criteria:

1. Intracranial hemorrhage is indicated on CT or MRI (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural or epidural hematoma).
2. History of intracranial hemorrhage; severe head trauma or stroke within the last 3 months.
3. Intracranial tumors, giant intracranial aneurysms.
4. Intracranial or spinal surgery within the last 3 months; major surgery within the last 2 weeks; arterial puncture at a site not easily compressed for hemostasis within the last 7 days.
5. Gastrointestinal or urinary system bleeding within the last 3 weeks.
6. Aortic dissection.
7. Acute bleeding tendency, including platelet count < 100×10^9/L or other bleeding tendencies.
8. Received low-molecular-weight heparin orally within 24 hours; taking warfarin with INR > 1.7 or PT > 15 seconds; used a new oral anticoagulant within 48 hours.
9. Blood glucose < 2.8 mmol/L or > 22.2 mmol/L.
10. Large area cerebral infarction indicated on head CT or MRI (infarction area > 1/3 of the middle cerebral artery territory).
11. Active visceral hemorrhage, known bleeding diathesis or significant bleeding disorders within the past 6 months
12. Severe ischemic stroke (NIHSS score > 25)
13. Epileptic seizures at the time of stroke onset
14. Pregnant or lactating women
15. Various terminal diseases with an expected survival of ≤ 3 months
16. Any other physical conditions where the doctor deems participation in this study may be detrimental to the patient
17. Currently participating in other drug or device clinical trials
18. mRS score > 2 before onset of the disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-08-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of symptomatic intracranial hemorrhage | Day 1
  The proportion of symptomatic intracranial hemorrhage within 24 hours after thrombolysis according to ECASS III criteria

SECONDARY OUTCOMES:
The proportion of symptomatic intracranial hemorrhage within 24 hours | DAY 1
  The proportion of symptomatic intracranial hemorrhage within 24 hours after thrombolysis (ECASS II criteria, SIST-MOST criteria, NINDS criteria)
The proportion of intracranial hemorrhage transformation | Day 1
  The proportion of any intracranial hemorrhage transformation within 24 hours after thrombolysis
The proportion of major substantive hemorrhage | The proportion of major substantive hemorrhage occurring within 24 hours after thrombolysis (PH2)
The proportion of severe or life-threatening major hemorrhage | DAY 90
  The proportion of severe or life-threatening major bleeding (as defined by GUSTO)
time to use of reperfusion treatment | DAY 1
  Door-to-needle time for intravenous thrombolysis patients
level of physical function | DAY 90
  Level of function defined across 7 categories of disability on the modified Rankin scale （mRS 0-6) in which scores of 0 or 1 indicate good function without or with symptoms but not disability, socress of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
death or dependency measured by a shift in mRS | DAY 90
  Level of function defined across 7 categories of disability on the modified Rankin scale （mRS 0-6) in which scores of 0 or 1 indicate good function without or with symptoms but not disability, socress of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Death | DAY 90
Neurological function measured by NIHSS | day 7 or at discharge
  NIHSS score at 7 days or at discharge (if the length of hospital stay is less than 7 days)
Neurological function measured by mRS | DAY 7 or at discharge
  mRS score at 7 days or at discharge (if the length of hospital stay is less than 7 days)
number of patients with serious adverse events | DAY 90
  total number of serious adverse events reported during follow-up, according to standard definitions

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with bona fide researchers after 1 year following conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after conclusion of the study